CLINICAL TRIAL: NCT07277842
Title: A Multicenter, Prospective, Phase III Randomized Controlled Trial of PD-1 Antibody Plus FOLFOXIRI Combined With Radiotherapy Versus CAPOX Combined With Radiotherapy as Total Neoadjuvant Therapy for pMMR Locally Advanced Low Rectal Cancer
Brief Title: PD-1 + FOLFOXIRI vs CAPOX as Total Neoadjuvant Therapy for pMMR Low Rectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHI-ZHONG PAN, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-302
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Low Rectal Adenocarcinoma; pMMR (Microsatellite Stable Rectal Cancer)
Keywords: pMMR locally advanced rectal cancer; total neoadjuvant therapy; PD-1 antibody; serplulimab; watch-and-wait
MeSH Terms: interventions — spartalizumab; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Serplulimab + FOLFOXIRI + Radiotherapy (Experimental): Participants in this arm will receive a PD-1 antibody (serplulimab) in combination with FOLFOXIRI chemotherapy and long-course pelvic radiotherapy as total neoadjuvant therapy before surgery. Treatment will be given according to the study protocol, with regular safety monitoring and response assessments.
  Interventions: Drug: Serplulimab; Drug: FOLFOXIRI chemotherapy; Radiation: Long-course pelvic radiotherapy
- Active Comparator: CAPOX + Radiotherapy (Active Comparator): Participants in this arm will receive CAPOX chemotherapy and long-course pelvic radiotherapy as total neoadjuvant therapy before surgery. Treatment will be given according to the study protocol, with regular safety monitoring and response assessments.
  Interventions: Drug: CAPOX chemotherapy; Radiation: Long-course pelvic radiotherapy

INTERVENTIONS:
Drug: Serplulimab — Serplulimab will be administered intravenously in combination with FOLFOXIRI chemotherapy and long-course pelvic radiotherapy as part of total neoadjuvant therapy in the experimental arm.
  Other Names: PD-1 antibody
  Arms: Experimental: Serplulimab + FOLFOXIRI + Radiotherapy
Drug: FOLFOXIRI chemotherapy — The FOLFOXIRI chemotherapy regimen (5-fluorouracil, leucovorin, oxaliplatin, irinotecan) will be administered according to the study protocol as part of total neoadjuvant therapy in the experimental arm, in combination with serplulimab and long-course pelvic radiotherapy.
  Other Names: 5-fluorouracil, leucovorin, oxaliplatin, irinotecan
  Arms: Experimental: Serplulimab + FOLFOXIRI + Radiotherapy
Drug: CAPOX chemotherapy — The CAPOX chemotherapy regimen (capecitabine plus oxaliplatin) will be administered according to the study protocol as part of total neoadjuvant therapy in the active comparator arm, in combination with long-course pelvic radiotherapy.
  Other Names: Capecitabine plus oxaliplatin
  Arms: Active Comparator: CAPOX + Radiotherapy
Radiation: Long-course pelvic radiotherapy — Long-course pelvic external beam radiotherapy will be delivered according to institutional standards as part of total neoadjuvant therapy in both study arms, in combination with chemotherapy (FOLFOXIRI plus serplulimab in the experimental arm or CAPOX in the active comparator arm).
  Other Names: External beam radiotherapy; Pelvic radiotherapy

SUMMARY:
The goal of this clinical trial is to find out if adding a PD-1 antibody (serplulimab) to FOLFOXIRI chemotherapy and radiotherapy works better than CAPOX chemotherapy with radiotherapy as total neoadjuvant therapy for adults with pMMR locally advanced low rectal cancer. It will also look at the safety of these treatments and how they affect long-term outcomes such as organ preservation and survival.

The main questions it aims to answer are:

Does PD-1 antibody plus FOLFOXIRI with radiotherapy improve 3-year event-free survival compared with CAPOX with radiotherapy?

Does this treatment increase the chance of clinical complete response and avoiding a permanent stoma (sphincter-preserving or non-surgical "watch-and-wait" management)?

What side effects and medical problems occur during and after these treatments?

Researchers will compare:

Group A (experimental group): PD-1 antibody (serplulimab) plus FOLFOXIRI chemotherapy combined with long-course radiotherapy as total neoadjuvant therapy.

Group B (control group): CAPOX chemotherapy combined with long-course radiotherapy as total neoadjuvant therapy.

Participants will:

Sign an informed consent form and have screening tests (physical exam, blood tests, ECG, imaging such as MRI/CT, endoscopy) to confirm they can join the trial.

Be randomly assigned (like drawing lots) to Group A or Group B. Receive several cycles of chemotherapy together with a 5-week course of pelvic radiotherapy before surgery; the experimental group will also receive PD-1 antibody during part of the chemotherapy and radiotherapy period.

Have regular clinic visits for checkups, blood tests, and assessment of side effects during treatment.

After neoadjuvant therapy, have MRI/CT and endoscopy to assess tumor response. Depending on the response, they may:

Receive surgery to remove the rectal tumor, or

If a clinical complete response is achieved and both doctor and patient agree, enter a "watch-and-wait" program instead of immediate surgery.

Provide blood samples and allow tumor tissue to be collected (for example, from biopsy and surgery) for future research (such as building PDX models and testing blood markers).

Be followed regularly for at least 5 years with clinic visits, blood tests (including CEA), imaging, and colonoscopy to check for tumor recurrence, side effects, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma.
* pMMR status documented by immunohistochemistry (MSH1, MSH2, MSH6 and PMS2 all positive) or by MSI testing showing MSS or MSI-L.
* Primary tumor located within 5 cm from the anal verge on pelvic MRI.
* Clinical stage cT3-4bN0M0 or cTxN+M0, with or without positive mesorectal fascia (MRF) and/or extramural vascular invasion (EMVI), and assessed by the multidisciplinary team as resectable with the potential for R0 resection.
* No clinical or radiologic evidence of bowel obstruction.
* No prior colorectal surgery.
* No prior chemotherapy or radiotherapy.
* No prior treatment with biologic agents (e.g., monoclonal antibodies), immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4), or other investigational drugs.
* Age 18 to 75 years (inclusive).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Estimated life expectancy > 2 years.
* Adequate bone marrow function: WBC > 3.5 × 10^9/L; platelets > 100 × 10^9/L; hemoglobin > 80 g/L.
* Adequate liver function: ALT and AST ≤ 1.5 × upper limit of normal (ULN); total bilirubin < 23.0 μmol/L.
* Adequate renal function: eGFR ≥ 60 mL/min/1.73 m² (CKD-EPI) or creatinine clearance (Ccr) ≥ 60 mL/min.
* Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

* Evidence of inguinal or lateral pelvic lymph node metastasis (lymph node short-axis diameter ≥ 7 mm or MRI features typical for metastatic lymph nodes).
* Clinically significant cardiac disease, including arrhythmias requiring anti-arrhythmic treatment (except β-blockers or digoxin), symptomatic coronary artery disease or myocardial ischemia (myocardial infarction within the last 6 months), or congestive heart failure > NYHA class II.
* Uncontrolled severe hypertension.
* History of HIV infection or active chronic hepatitis B (HBV DNA > 2 × 10^3 IU/mL) or hepatitis C (HCV RNA > 1 × 10^3 IU/mL).
* Active pulmonary tuberculosis under treatment or having received anti-tuberculosis therapy within 1 year before screening.
* Other active severe infections (as defined by NCI-CTCAE v5.0).
* Evidence of distant metastasis outside the pelvis before treatment.
* Cachexia or decompensated organ dysfunction.
* Prior pelvic or abdominal radiotherapy.
* Multiple primary colorectal cancers.
* History of seizures requiring ongoing treatment (e.g., corticosteroids or anti-epileptic drugs).
* History of another malignancy within the past 5 years, except adequately treated cervical carcinoma in situ or basal cell carcinoma of the skin.
* Drug or alcohol abuse, or any medical, psychological, or social condition that, in the investigator's judgment, could interfere with study participation or the evaluation of study results.
* Any active autoimmune disease or history of autoimmune disease (including but not limited to interstitial pneumonia, uveitis, colitis, hepatitis, hypophysitis, nephritis, hyperthyroidism, or hypothyroidism).
* Receipt of any prophylactic vaccine against infectious diseases (e.g., influenza, varicella) within 4 weeks before enrollment.
* Requirement for long-term immunosuppressive therapy or systemic/local corticosteroids at immunosuppressive doses (equivalent to > 10 mg/day of prednisone or other corticosteroids).
* Known or suspected allergy or hypersensitivity to any study drug or to any component of the study treatments.
* Any unstable condition or other circumstance that may, in the opinion of the investigator, compromise patient safety or study compliance.
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling or unable to use adequate contraception during the study.
* Refusal or inability to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2028-12-29 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
3-year Event-Free Survival (EFS) | Up to 3 years after randomization
  Event-free survival (EFS) is defined as the time from randomization to the first occurrence of any of the following events: (1) locoregional failure, including unresectable primary tumor after completion of total neoadjuvant therapy, R2 resection (macroscopic residual tumor), or local bed recurrence after R0-R1 resection; (2) distant metastasis; (3) new invasive primary colorectal cancer; or (4) death from any cause. Patients without an event at the time of analysis will be censored at the date of the last tumor assessment.

SECONDARY OUTCOMES:
Clinical Complete Response (cCR) Rate | At 10-14 weeks after completion of radiotherapy (response assessment prior to definitive management)
  Proportion of participants achieving clinical complete response (cCR) after completion of total neoadjuvant therapy. cCR will be assessed by digital rectal examination, endoscopy, pelvic MRI and serum CEA according to predefined criteria (no palpable tumor, endoscopic whitening or telangiectasia only, fibrotic signal on MRI without residual tumor or nodes, and normal CEA).
Anal Sphincter Preservation Rate | From randomization to definitive management (surgery or decision for watch-and-wait) and last follow-up, up to approximately 1 year after randomization
  Proportion of participants who achieve anal sphincter preservation, defined as undergoing sphincter-preserving surgery (e.g., low anterior resection, intersphincteric resection) or managed with a watch-and-wait strategy without permanent stoma at last follow-up.
Incidence of Treatment-related Adverse Events During Total Neoadjuvant Therapy | From first dose of study treatment until 30-90 days after completion of chemotherapy/radiotherapy or surgery, up to approximately 1 year after randomization
  Number and proportion of participants experiencing treatment-related adverse events during total neoadjuvant therapy, graded according to NCI-CTCAE version 5.0. Both overall adverse events and grade 3-5 toxicities related to chemotherapy, immunotherapy, or radiotherapy will be summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: No